CLINICAL TRIAL: NCT01954134
Title: P53 Antibody; Is it an Indicator of Dedifferentiated Thyroid Cancer?
Brief Title: P53 in Differentiated Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Zekiye HASBEK, M.D., Assistant Professor, Cumhuriyet University, School of Medicine, Department of Nuclear Medicine, Cumhuriyet University
Other Study IDs: T-485; T-485 (Other: Cumhuriyet University Scientific Research Project Unit)
Record Dates: First submitted 2013-09-11; First posted 2013-10-01 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Thyroid Neoplasms
Keywords: Tumor Suppressor Protein p53,; Iodine Radioisotopes
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- thyroid cancer, healty: Thyroid cancer group: patients with differentiated or dedifferentiated thyroid cancer Healty: control group

SUMMARY:
In clinical practise patients with negative radioiodine scan with positive tyhroglobulin is considered as radioiodine resistant or in another words in the process of dedifferentiation. The aim of the present study was to search a simple blood test that could lead to early identification of patients with dedifferentiation. In this respect, we investigate whether the serum level of anti-p53 antibody has the diagnostic value in the follow-up of patients with high levels of thyroglobulin (tg) and negative I-131 scan.

DETAILED DESCRIPTION:
In the present study enrolled were 171 patients with mean age of 47.7±13.5 yrs (range; 16-80yrs) and 28 healthy subjects with an age range of 18-52 yrs (mean: 36.0±9.8 yrs). 134 (78.4%) patients were female and 37 (21.6%) patients were male.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with DTC
* Treated with total and/or near-total thyroidectomy
* Referred for I-131 ablation therapy or low dose I-131 whole body scan (WBS)
* Between December 2010 and January 2013.

Exclusion Criteria:

* Dose 131-I given in another hospital
* Radioiodine treatment more than one year after thyroidectomy.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 171 patients with an age range of 16-80 yrs (mean: 47.7±13.5 yrs) and a total of 28 healthy subjects with an age range of 18-52 yrs (mean: 36.0±9.8 yrs) were included in this study.
Sampling Method: Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2010-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
There was not any risk for patients. | with in the first 8-10 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zekiye Hasbek, M.D., Principal Investigator — Cumhuriyet University
Locations (1):
- Cumhuriyet University, School of Medicine, Dept. of Nuclear Medicine, Sivas, Turkey (Türkiye)

REFERENCES:
- [Result] Wu M, Mao C, Chen Q, Cu XW, Zhang WS. Serum p53 protein and anti-p53 antibodies are associated with increased cancer risk: a case-control study of 569 patients and 879 healthy controls. Mol Biol Rep. 2010 Jan;37(1):339-43. doi: 10.1007/s11033-009-9744-7. Epub 2009 Aug 20. PMID 19693693
- [Result] Muller M, Meyer M, Schilling T, Ulsperger E, Lehnert T, Zentgraf H, Stremmel W, Volkmann M, Galle PR. Testing for anti-p53 antibodies increases the diagnostic sensitivity of conventional tumor markers. Int J Oncol. 2006 Oct;29(4):973-80. PMID 16964393
- [Derived] Hasbek Z, Turgut B, Erselcan T. p53 antibody: is it an indicator of dedifferentiated thyroid cancer? Ann Nucl Med. 2014 Jan;28(1):42-6. doi: 10.1007/s12149-013-0783-8. PMID 24234516